CLINICAL TRIAL: NCT05324852
Title: AGItated Patients Management: intraNASAL Midazolam vs Intramuscular Loxapine, a Randomized Non Inferiority Trial
Brief Title: AGItated Patients Management: intraNASAL Midazolam vs Intramuscular Loxapine
Acronym: AGINASAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision:
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Lariboisière-Saint Louis clinical research unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160947J
Record Dates: First submitted 2022-03-21; First posted 2022-04-12 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Midazolam; Loxapine

STUDY DESIGN:
Intervention Model Description: Intramuscular loxapine versus intranasal midazolam
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal midazolam (Experimental): Midazolam, 5 mg, injectable solution in 5mg/ml, if weight < 50 kg : 5mg; if weight ≥50kg : 10mg, intranasal administration, atomize into nose with Mucosal Atomizer Device (MAD) 5mg(1ml) up each nostril , one time
  Interventions: Drug: Intranasal midazolam
- Intramuscular loxapine (Active Comparator): Loxapine, 100mg, injectable solution in 50mg/2ml intramuscular, intra muscular administration, one time
  Interventions: Drug: Intramuscular loxapine

INTERVENTIONS:
Drug: Intranasal midazolam — Midazolam, 5 mg, injectable solution in 5mg/ml, intranasal administration, atomize into nose with Mucosal Atomizer Device (MAD) 5mg(1ml) up each nostril , one time
  Other Names: Midazolam
  Arms: Intranasal midazolam
Drug: Intramuscular loxapine — Loxapine, 100mg, injectable solution in 50mg/2ml intramuscular, intra muscular administration, one time
  Other Names: Loxapine
  Arms: Intramuscular loxapine

SUMMARY:
This study is a non-inferiority phase III randomized trial evaluating the effect of intranasal midazolam versus intramuscular loxapine on the rapid tranquilization of agitated patient in emergency department. Intranasal midazolam is safe and may allow a management of extreme agitation state and prevent adverse effects.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label randomized, controlled, parallel-group 2-arm phase III non-inferiority trial. Patients with agitation at emergency department will be randomized to two arms of treatment: one experimental arm with intranasal midazolam 5mg (investigational medicinal product), and one control arm with comparator treatment intramuscular loxapine 100mg. The duration of participation for each patient is at least 28 days (+7 days if follow-up not completed on D28). An endpoint Adjudication Committee will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years;
* Agitated Patient whose somatic or psychiatric aetiology cannot be diagnosed in an emergency situation and who need a sedation in a hospital emergency setting due to the presence of unmanageable agitation with 3 major criteria.

Major criteria :

Agitation Pain Tolerance Tachypnea ( fr > 20)

And 1 minor criteria among :

Sweating Tactile Hyperthermia Medical care Non compliance Lack of tiring Unusual Strenght Inappropriately clothed, nudity

• Medical insurance The protocol can start if the THREE major inclusion criteria and ONE of the minor inclusion criteria are checked PRESENT and ALL the non-inclusion criteria are checked no.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from randomization into the study:

* Pregnancy
* Prisoners
* Contraindications to intranasal Midazolam or intramuscular Loxapine :

  * Hypersensitivity to benzodiazepines or to any of the excipients (Sodium Chloride, Hydrochloric Acid, Sodium Hydroxide, Water for Injection)
  * Known hypersensitivity to loxapine or to any of the excipients (Polysorbate 80, propylene glycol, 20% v/v hydrochloric acid, water for injections, Nitrogen (Inert gas)
  * Individuals who are in comatose states or have central nervous system (CNS) depression due to alcohol or are taking other depressant drugs
  * Individuals with severe depressive states, spastic diseases, and with Parkinson's disease, except in the case of dyskinesias due to levodopa treatment
  * In combination with dopamine agonists except levodopa (amantadine, bromocriptine, lisuride, pergolide, piribedil, ropinirole, cabergoline, pramipexole, apomorphine) outside the patient with Parkinson's disease
  * Individuals with a history of cerebrovascular accident or epilepsia
  * Individuals in whom a significant elevation of blood pressure would constitute a serious hazard, such as patients with significant hypertension;
  * Individuals with severe cardiac decompensation
  * Patients with severe respiratory failure or acute respiratory depression
  * Individuals with acute narrow angle glaucoma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2023-04-09 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Evolution of agitation | 15 minutes
  The proportion of patients with sufficient improvement of agitation at 15 minutes defined by a reduction of at least 3 points on the CGI (Clinical Global Impression).

SECONDARY OUTCOMES:
Incidence of adverse events following the use of loxapine or midazolam | 240 minutes
  The adverse effects over 240 minutes : oxygen desaturation [<90%], airway obstruction requiring intervention, tracheal intubation, cardiac arrhythmias, prolonged QTc interval, hypotension, extrapyramidal side effects, akathisia, and anaphylaxis.
Number of deceased patients | 24 hours
  mortality at 24 hours
Number, type and severity level of adverse events | 240 minutes
  The adverse effects over 240 minutes : oxygen desaturation [<90%], airway obstruction requiring intervention, tracheal intubation, cardiac arrhythmias, prolonged QTc interval, hypotension, extrapyramidal side effects, akathisia, and anaphylaxis
level of sedation obtained by loxapine or midazolam. | 15,60,120 and 240 minutes
  The proportion of patients with sufficient improvement of agitation at 240 minutes defined by a reduction of at least 3 points on the CGI.
  Proportion of patients clinically improved on the improvement subscale of the clinical global impressions scale at 15, 60, 120, and 240 minutes.
level of sedation obtained by loxapine or midazolam. | 15 minutes
  Proportion of patients with additional sedation required
feelings of health providers with Qualitative research. | 15 min and 240 min
  Duration of violent and acute behavioural disturbance Staff injuries. Proportion of patients requiring the doctor to be called back.
Improvement of agitation | 15 min
  The proportion of patients with sufficient improvement of agitation at 15 minutes defined by a RASS < -1

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Adnet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No